CLINICAL TRIAL: NCT02915107
Title: Randomized Comparison of Vascular Healing of a Polymer-Free Biolimus-eluting BIOFREEDOM Stent With a Biodegradable-Polymer Sirolimus-eluting ORSIRO Stent in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: The SORT OUT IX STEMI OCT Trial
Acronym: OCT STEMI SOIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lisette Okkels Jensen, MD DMSci, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SO IX OCT STEMI
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Acute Myocardial Infarction
Keywords: drug eluting stents; coronary vascular healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biofreedom (Experimental): Experimental: Biofreedom BioFreedom stent at index procedure
  Interventions: Device: BioFreedom
- Orsiro (Active Comparator): Active comparator: Orsiro Orsiro stent at index procedure
  Interventions: Device: Orsiro

INTERVENTIONS:
Device: BioFreedom — PCI with BioFreedom
  Arms: Biofreedom
Device: Orsiro — PCI with BioFreedom
  Arms: Orsiro

SUMMARY:
The aim of the Danish Organization for Randomized Trials with Clinical Outcome (SORT OUT) IX STEMI OCT is to compare early vascular healing of the polymer-free Biolimus-eluting BIOFREEDOM stent with a biodegradable-polymer Sirolimus-eluting ORSIRO stent in patients with ST-segment elevation myocardial infarction (STEMI) treated with primary percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
SORT OUT IX STEMI OCT is a randomized 1:1 study comparing the polymer-free Biolimus-eluting BIOFREEDOM stent with a biodegradable-polymer Sirolimus-eluting ORSIRO stent patients with STEMI treated with primary PCI.

Vascular healing index (uncovered stent struts, malapposed stent struts, maximal intima coverage and accumulated extra-stent lumen volume) assessed with optical coherence tomography (OCT) 1 month after primary PCI.

Patients will be enrolled by the investigators and randomly allocated to treatment groups after diagnostic coronary angiography and before primary PCI. A web based Trial Partner randomization system will be used.

OCT will be performed with the frequency-domain OPTIS OCT system and Dragonfly™ Imaging Catheter during the index procedure and after 1 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or over with STEMI, requiring treatment with a drug-eluting stent.

Exclusion Criteria:

* life expectancy of less than one year; an allergy to aspirin, clopidogrel, ticagrelor, prasugral, biolimus or sirolimus; participation in another randomized trial; chronic renal disease; or inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Vascular healing index (uncovered stent struts, malapposed stent struts, maximal intima coverage and accumulated extra-stent lumen volume) assessed with optical coherence tomography (OCT) 1 month after primary PCI. | Primary endpoint assessed after 1 month

SECONDARY OUTCOMES:
Target lesion failure | 1 year, 2 years, 3 years, 4 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisette Okkels Jensen, MD DMSci PhD, Principal Investigator — Odense University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital, Copenhagen
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Hansen KN, Maeng M, Antonsen L, Maehara A, Jakobsen L, Ellert J, Terkelsen CJ, Ahlehoff O, Thim T, Fallesen CO, Noori M, Veien KT, Jensen LO, Christiansen EH. Early vascular healing after implantation of the polymer-free biolimus-eluting stent or the ultrathin strut biodegradable polymer sirolimus-eluting stent in patients with ST-segment elevation myocardial infarction. Coron Artery Dis. 2022 May 1;33(3):196-205. doi: 10.1097/MCA.0000000000001113. PMID 34985003